CLINICAL TRIAL: NCT05093400
Title: Oropharynx (OPX) Salivary Biomarker Study: Microbiome, Virome, and Metabolomics
Brief Title: Oropharynx (OPX) Salivary Biomarker Study
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Kathryn (Katie) M. Van Abel, Principal Investigator, Mayo Clinic
Other Study IDs: 21-006529
Record Dates: First submitted 2021-09-17; First posted 2021-10-26 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Blood, saliva, and tumor tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Normal Saliva: saliva from "normal healthy" adults.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — saliva collection

SUMMARY:
The goal of this study is to analyze certain biomarkers to look at the relationship between HPV in the saliva, stage at presentation, and a potential self-test compared to saliva of non-cancerous participants.

ELIGIBILITY:
Inclusion Criteria:

* Oropharynx or Oral Cavity Squamous Cell Carcinoma Patients: collected under the OPX Biomarker Protocol (IRB: 19-006036).

Normal Controls:

* Age ≥ 18 years;
* Able to provide informed written consent documenting permission to give saliva sample for research testing.;
* Ability to complete questionnaire(s) by themselves or with assistance.

Exclusion Criteria:

* Oropharynx or Oral Cavity Squamous Cell Carcinoma Patients: collected under the OPX Biomarker Protocol (IRB: 19-006036).

Normal Controls:

* Any personal history of head or neck cancer including head or neck skin cancer.
* Other active malignancy ≤ 5 years prior to registration.
* EXCEPTIONS: Non-melanotic skin cancer, non-metastatic prostate cancer.
* NOTE: If there is a history of prior malignancy, they must not be receiving other specific treatment for their cancer.
* Dry mouth (xerostomia) caused by any chronic (>30 days) condition (known or unknown) or medication.
* Recent (within 30 days) or active upper aerodigestive tract or anogenital infections.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy non-cancerous participants
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-09-17 (Actual); Primary Completion 2023-05-02 (Actual); Study Completion 2023-05-05 (Actual)

PRIMARY OUTCOMES:
Oncologic strains in HPV DNA salivary samples | 2 years
  Number of patients to have oncologic strains of HPV DNA in salivary samples

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Van Abel, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials